CLINICAL TRIAL: NCT04939064
Title: Endometrial Basis for Infertility in Women With Recurrent Implantation Failure and Pregnancy Loss
Status: Terminated | Type: Observational
Why Stopped: lapse in approval
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000206; 000206-CH
Record Dates: First submitted 2021-06-24; First posted 2021-06-25 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Normal Endometrial Physiology
Keywords: IVF; RPL; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ART Infertile: Women that are part of a couple diagnosed with unexplained infertility that conceived on the first embryo transfer (ET) attempt
- Early Implantation Failure (EIF): Infertility defined by a failure to conceive after: a) three or more failed transfers of high-quality blastocyst(s) (grade 3BB or higher); or b) two or more transfers of euploid blastocyst
- Early Pregnancy Failure (EPF): defined by two or more biochemical pregnancies after transfer of a high-quality or euploid blastocyst with a positive hCG 12 days after ET but without subsequent clinical signs of pregnancy
- Normal Fertile: Women with proven parity based on spontaneous conception without fertility treatment or prior diagnosis of infertility, normal uncomplicated pregnancy, birth of at least one healthy baby
- Recurrent Pregnancy Loss (RPL): defined as the loss of two or more pregnancies after transfer of a high-quality or euploid blastocyst with a positive HCG 12 days after ET and subsequent clinical signs of pregnancy

SUMMARY:
Background:

Pregnancy loss is the most common complication of pregnancy. It occurs in roughly one-half

of natural conceptions. It most frequently occurs in the first 2 to 3 weeks of pregnancy. Researchers want to look at the lining of the uterus, called the endometrium, to see what role it plays in implantation and miscarriage.

Objective:

To gain a better understanding of how normal and abnormal endometrium works.

Eligibility:

Healthy, fertile women ages 18-42 who have had one prior child.

Design:

Participants will have 3 study visits.

At visit 1, participants will have a medical history. They will have a radiologic/imaging review if needed. They will be taught how to monitor their urine luteinizing hormone (LH) at home with an ovulation predictor kit. They will have their second study visit 9 days after their LH surge.

At visit 2, participants will take a urine pregnancy test. They will have a physical exam and have blood drawn. They will have a uterine lavage and endometrial biopsy. For this, a speculum will be placed into the vagina. A soft catheter will be inserted through the cervical canal into the uterus. Saline will be added into the uterus and then recovered after 30 seconds. A tissue sample will be taken.

About 46 days later, participants will start another round of LH monitoring. They will have a third study visit 9 days after their LH surge. At visit 3, they will repeat the tests from visit 2.

Some samples will be used for genetic tests.

Participation will last for 3 menstrual cycles.

...

DETAILED DESCRIPTION:
Pregnancy loss is the most common complication of human gestation, occurring in roughly one-half of natural conceptions and most frequently in the first two to three weeks of gestation. In recent years it has become apparent that constitutive endometrial dysfunction represents an important contributor to infertility in women being treated with assisted reproductive technologies (ART). This application is specifically focused on the endometrial origins and basis of embryo implantation failure (EIF), early pregnancy failure (EPF), and recurrent pregnancy loss (RPL) in ART patients. The central hypothesis is that idiopathic infertility primarily stems from constitutive endometrial dysfunction, attributable to defects in progesterone responsiveness of the endometrial epithelium and stroma as well as immune cells. The goal of this research is to begin testing this hypothesis by focusing on infertile women experiencing the continuum of first trimester pregnancy loss. A team of exceptional extramural and intramural investigators with complementary and substantial expertise in basic reproductive biology and translational reproductive sciences will address that hypothesis by conducting a collaborative research project. At the NIH Clinical Center, the endometrium from cohorts of normal healthy fertile donors and infertile patients with carefully phenotyped and clinically-defined EIF, EPL or RPL will be biopsied in an outpatient setting (Aim 1). Advanced single cell technologies will be used to interrogate the endometrium (Aim 1). Organoids will be used to functionally study progesterone responses of the endometrial epithelium (Aim 2). In vitro decidualization will be used to functionally interrogate hormone responsiveness and decidualization capacity of the endometrial stroma and understand the influence of decidual immune cells (Aim 3). Cutting-edge genomic and transcriptomic technologies and advanced bioinformatics and data integration will be used to understand cell type heterogeneity, cell-specific differences in gene expression, and discern critical progesterone-driven biological pathways important for endometrial function that are disrupted in infertile women. The proposed aims are conceptually and technically innovative and together will have a broad impact on the field by filling a substantial gap in our fundamental knowledge of uterine biology and infertility. This application specifically targets NIH funding opportunity announcement PAR-18-951 entitled Opportunities for Collaborative Research at the NIH Clinical Center and focuses on major research priorities of the Fertility and Infertility Branch of the NICHD. These efforts will contribute to our understanding of the cellular basis of idiopathic infertility, enable the development of new tests enabling clinicians to diagnose and prescribe regimens directed at treating specific underlying endometrial dysfunction, and ultimately impact pregnancy outcomes in assisted and natural conceptions enabled by a personalized medicine approach.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Female, aged 18-42, childbearing potential
* In good general health as evidenced by medical history, previous fertility or diagnosed with infertility with and without a previous pregnancy loss.

  * Normal Fertile - Control- Women with proven parity based on spontaneous conception without fertility treatment or prior diagnosis of infertility, normal uncomplicated pregnancy, and birth of at least one healthy baby
  * ART Infertile - Control-Women that are part of a couple diagnosed with unexplained infertility that conceived on the first embryo transfer (ET) attempt and meet inclusion/exclusion criteria.
  * Early Implantation Failure (EIF) - Infertility defined by a failure to conceive after:

    a) three or more failed transfers of high-quality blastocyst(s) (grade 3BB or higher); or b) two or more transfers of euploid blastocyst(s) (tested through trophectoderm biopsy and preimplantation genetic testing for aneuploidy (PGT- A) using next generation sequencing). These women will have a negative serum beta human chorionic gonadotropin (hCG) 12 days after ET.
  * Early Pregnancy Failure (EPF) - Infertility defined by two or more biochemical pregnancies after transfer of a high-quality or euploid blastocyst with a positive hCG 12 days after ET but without subsequent clinical signs of pregnancy (detection of intrauterine or extrauterine gestational sac at 5-7 weeks of gestation). While, by definition these are pregnancies of unknown location (PUL) and will

include spontaneously resolving ectopic pregnancies, the vast majority of these will be failed intrauterine pregnancies.

--Recurrent Pregnancy Loss (RPL): Infertility defined by the loss of two or more pregnancies after transfer of a high-quality or euploid blastocyst with a positive HCG 12 days after ET and subsequent clinical signs of pregnancy (detection of an intrauterine gestational sac at 5-7 weeks gestation by ultrasound).

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Women with prior hysterectomy as they do not have an endometrium
* Postmenopausal women
* Women with a history of preterm delivery (<37-week gestation), preeclampsia and/or stillbirth are excluded.
* Women with RPL must screen negative for the antiphospholipid syndrome (negative lupus anticoagulant, negative IgG and IgM antiphospholipid antibodies and negative IgG and IgM anti-2GP1 antibodies)
* Women suffering from infertility with and without early pregnancy loss with prior diagnosis of common known disease risk factors, including disorders such as uterine anomalies, coagulopathy, balanced translocation, gynecological disease, other reproductive disorders and/or autoimmune conditions, pathology confirmed or suspected endometriosis, pathology confirmed or suspected adenomyosis, endometrial polyp(s) or submucosal fibroids, pathology confirmed acute or chronic endometritis, hydrosalpinx communicating with the endometrial cavity, history of Asherman syndrome, poorly controlled endocrinopathies, HIV infection, ovarian insufficiency and irregular menstrual cycles
* Women who are currently Pregnant as we would not be able to obtain an endometrial sample
* History of gonadotoxic therapy, precancerous (endometrial hyperplasia) or cancerous condition of the female reproductive tract,
* Current smoker or tobacco use or tobacco use within 30 days.
* Current use of reproductive hormones and/or fertility medications
* Current use of steroids or non-steroidal anti-inflammatory agents within the last 3 days.
* Women who are obese (BMI >30)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The gynecological populations at both NIH Clinical Centers and WRNMMC are 46% Caucasian, 20% African American, 25% Hispanic, 5% Asian, and 4% other. Patients consist of military women or their families and patients enrolled in studies at the NIH.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Single cell analysis of the endometrium from fertile and infertile women. | 7-9 days post LH surge in cycling women
  This aim hypothesizes that the endometrium of fertile women has intrinsic differences in cell types and cell-specific gene expression compared to infertile women with clinically-defined early pregnancy loss. Cohorts of fertile women (controls) and infertile women with EIF, EPF or RPL (cases) will be recruited and sampled. Endometrial biopsies will be obtained from the women during the mid-secretory phase (LH+7-9) of their cycle. Single nuclei RNA-seq (snRNA-seq) will be employed to define the transcriptomes of all cells in the endometrial biopsies. Immunohistochemical analysis of an epithelial receptivity marker (FOXO1) and advanced bioinformatics analysis will provide a detailed understanding of cell heterogeneity and cell type-specific differences in gene expression in the endometrium of fertile and infertile women.

SECONDARY OUTCOMES:
Understanding endometrial epithelial cell response to progesterone using organoids | in patients with abnormal progesterone receptor signaling
  This aim hypothesizes that endometrium of infertile women has intrinsic defects in epithelial cell responses to progesterone (P4) compared to endometrium of fertile women via altered progesterone receptor and FOXO1 signaling, however only a subset of patients may have alterations in those pathways. Endometrial epithelial organoids (EEO) will be derived from the isolated epithelial cells of endometrial biopsies from Aim 1 using an established three-dimensional (3D) culture system. The responsiveness of the EEO to P4 will be interrogated using single cell RNA-seq, single cell ATAC-seq, and whole transcriptome (total bulk RNA-seq) analyses. Advanced bioinformatics analysis data will reveal cell type-specific and genomic differences in progesterone responsiveness of EEO underlying infertility in the case cohorts.
Understanding endometrial stromal cell response to progesterone and immune cells using in vitro decidualization. | after culture in IVD system
  This aim hypothesizes that endometrium of infertile women has intrinsic defects in SC decidualization due to P4 resistance and/or immune cell composition and responsiveness compared to endometrium of fertile women. Stromal cells and immune cells from the endometrial biopsies in Aim 1 will be isolated and cultured using an established in vitro decidualization (IVD) system. The ability of the SC to differentiate into functional and senescent DC in response to P4 without or with decidual immune cells will be determined by single cell and whole transcriptome analyses combined with advanced bioinformatics analysis. An integrative meta-analysis will be used to understand the cellular basis of idiopathic infertility, identify potential biomarkers of endometrial receptivity, fertility, and infertility, and discover novel pathways that can be used to develop personalized medicine treatments for idiopathic fertility and improve outcomes in assisted and natural pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Laverne G Mensah, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000206-CH.html